Official Title: Phase 2, Open-label, Multiple-dose Trial to Assess the Safety, Tolerability,

Pharmacokinetics, and Efficacy of Delamanid (OPC 67683) in Pediatric Multidrug-resistant Tuberculosis Patients on Therapy with an Optimized Background Regimen of Antituberculosis Drugs over a 6-Month

**Treatment Period** 

NCT Number: NCT01859923

**Document Date:** SAP Version Final: 03 July 2019



# Otsuka Pharmaceutical Development & Commercialization, Inc.

#### Investigational New Drug OPC-67683 (Delamanid)

Protocol No. 242-12-233

IND No. 76,728

Phase 2, Open-label, Multiple-dose Trial to Assess the Safety, Tolerability, Pharmacokinetics, and Efficacy of Delamanid (OPC 67683) in Pediatric Multidrug resistant Tuberculosis Patients on Therapy with an Optimized Background Regimen of Antituberculosis Drugs over a 6 Month Treatment Period

Investigational Medicinal Product Delamanid (OPC-67683)

# **Statistical Analysis Plan**

Version: Final Date: 3 July 2019

Protocol Version Amendment 5: 28 February 2019

Confidential

May not be used, divulged, published or otherwise disclosed without the consent of Otsuka Pharmaceutical Development & Commercialization, Inc.

# **Table of Contents**

| <b>Table</b> | of Contents | 2 |
|--------------|------------------------------------------|----|
| List of | In-text Tables | 4 |
| List of | In-text Figures | 5 |
| List of | Appendices | 6 |
| | Abbreviations and Definitions of Terms | |
| | ntroduction | |
| | tudy Objectives | |
| 2.1 | Primary Objectives | |
| 2.2 | Secondary objectives: | 9 |
| 3 S | tudy Design | 9 |
| 4 S | ample Size and Power Justification | 11 |
| 5 S | tatistical Analysis | 11 |
| 5.1 | General Principles | 11 |
| 5.2 | Datasets for Analysis | 12 |
| 5.3 | Definition of Baselines | 12 |
| 5.4 | Handling of Missing Data | 12 |
| 5.5 | Demographic and Baseline Characteristics | 12 |
| 5.6 | Medical History | 12 |
| 5.7 | Primary Outcome Analysis | 13 |
| 5.7.1 | Safety Outcome Variables | 13 |
| 5.7.1.1 | Adverse Events. | 13 |
| 5.7.1.2 | Clinical Laboratory Data | 14 |
| 5.7.1.3 | Drug Induced Liver Injury (DlLI) | 15 |
| 5.7.1.4 | Physical Examination and Vital Signs | 15 |
| 5.7.1.5 | Electrocardiogram Results | 15 |
| 5.7.1.6 | Additional Safety Assessments | 16 |
| 5.8 | Extent of Exposure to Trial Medication | 16 |
| 5.9 | Treatment Compliance | 16 |
| 5.10 | Protocol Deviation | 16 |

| 1 | P | r | _ | ٠ | t. | n | | ٠, | _ | J | ١٠ | | ) / | 1 | ) | _ | 1 | 2 | _ | 2 | 2 | , |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| ı | Г | | u | ) | и | o | u | 51 | u | ) | | - / | | + | 7. | - | | / | _ | • / | . 1 | ) |

| 7 | Bibliography | 28 |
|---|---|---|
| 6 | <b>Table of Contents for Table and Listings</b> | 20 |
| 5.15 | Discontinuation | 18 |
| 5.14 | Patient Disposition, Completion Rate and Reasons for Discontinuation | 18 |
| 5.13 | Concomitant Medications | 18 |
| 5.12.4 | Final Treatment Outcomes Assessed by the Principal Investigator | 18 |
| 5.12.3 | Palatibility | 18 |
| 5.12.2 | Efficacy Outcome Analysis | 17 |
| 5.12.1 | Pharmacokinetics/Phamacodynamics | 17 |
| 5.12 | Secondary Outcome Analysis | 17 |
| 5.11.1 | Pharmacokinetic Assessment of Cerebral Spinal Fluid (CSF) | 17 |
| 5.11 | Pharmacokinetic Analysis of Plasma | 16 |

| Table 3-1 | Subject Population |
|-----------|--------------------|
|-----------|--------------------|

| List of In-text Figu | ures |
|----------------------|------|
|----------------------|------|

| Figure 3-1 | Trial Design Schematic 1 | 1 |
|------------|--------------------------|---|
| _ | | |

# **List of Appendices**

| Appendix 1 | Serum Chemistry, Hematology and Urinalysis Lab Test<br>Results Clinical Significant Criteria Based on Division of<br>AIDS (DAIDS) Table for Grading the Severity of Adult and<br>Pediatric Adverse Events | 29 |
|---|---|---|
| Appendix 2 | Criteria for Potentially Clinical Significant Vital Sign<br>Abnormalities | 32 |
| Appendix 3 | Criteria for Potentially Clinical Significant ECG Abnormalities | 33 |

**IEC** 

**IMP** 

INH

#### List of Abbreviations and Definitions of Terms

Definition **Abbreviation** Adrenocorticotropic hormone ACTH Analysis data model **ADAM** Subject-level analysis dataset **ADSL** AΕ Adverse event Acid-fast bacilli AFB Acquired immunodeficiency syndrome **AIDS** ALT Alanine aminotransferase Activated partial thromboplastin time aPTT **ARV** Antiretroviral AST Aspartate aminotransferase ATC Anatomical Therapeutic Chemical Area under the plasma-time concentration curve **AUC** AUC0-24 Area under the plasma-time concentration curve from time zero to 24 hours Dosing twice per day BID Body mass index BMI Blood pressure BP Competent authority CA **CDISC** Clinical Data Interchange Standards Consortium **CFU** Colony Forming Units CI Confidence interval Peak (maximal) concentration of drug in plasma/serum Cmax Contract Research Organization **CRO** Cerebral Spinal Fluid CSF Cytochrome P-450 CYP Drug Induced Liver Injury DILI Directly-observed therapy short-course **DOTS** Drug susceptibility testing DST Drug-susceptible tuberculosis DS-TB EB Ethambutol Early bactericidal activity **EBA** Ethics committee EC Electrocardiogram ECG electronic case report form eCRF **EFV** Efavirenz European Union EU (United States) Food and Drug Administration FDA **FOCBP** Female of child-bearing potential Good Clinical Practice **GCP** HBsAg Hepatitis B surface antigen Hepatitis C virus **HCV** HIV Human immunodeficiency virus HR Heart rate Investigator's brochure IΒ Inhibitory concentration IC Informed consent form **ICF** ICH International Conference on Harmonization Identification ID Interval duration measurement **IDM** 

Statistical Analysis Plan 7 of 33 Version Date: 3 July 2019

**Independent Ethics Committee** 

Isoniazid

Investigational medicinal product

INR International normalized ratio IRB Institutional review board IRE Immediately reportable event ISR Immediate Safety Report LMP Last menstrual period

LPV Lopinavir

LTBI Latent TB infection

MedDRA Medical Dictionary for Regulatory Activities

MD Medical doctor

MDR-TB Multidrug-resistant tuberculosis
MTB Mycobacterium tuberculosis
NTBP National Tuberculosis Program
OBR Optimized background regimen

PD Pharmacodynamic P-gp P-glycoprotein

PIP Pediatric Investigational Plan

PK Pharmacokinetics

PO Oral route of administration POPPK Population pharmacokinetics

PT Preferred term
PZA Pyrazinamide
QD Once daily

QTc Corrected QT interval

QTcB QTc corrected by Bazett formula QTcF QTc corrected by Fridericia formula

RR Respiratory rate
RTV Ritonavir

SAE Serious adverse event SCC Sputum culture conversion

SD Standard deviation

SMC Safety Monitoring Committee

SOC System organ class TB Tuberculosis

TEAE Treatment-emergent adverse event

TFV tenofovir

t1/2 Elimination half-life

t1/2z Terminal elimination half-life TSH Thyroid stimulating hormone

TST Tuberculin skin test
ULN Upper limit of normal
WHO World Health Organization
XDR-TB Extensively Drug Resistant TB

#### 1 Introduction

This statistical analysis plan (SAP) documents the statistical methodology and data analysis algorithms and conventions to be applied for statistical analysis and reporting of safety, tolerability, pharmacokinetics (PK) and efficacy of Otsuka Pharmaceutical Development and Commercialization (Otsuka) Trial 242-12-233. All amendments to the protocol are taken into consideration in developing this SAP.

# 2 Study Objectives

# 2.1 Primary Objectives

- Safety and tolerability: To evaluate the long-term safety and tolerability of delamanid and its metabolites in combination with an OBR during a 6-month treatment period in pediatric patients with MDR-TB for the age-specific delamanid doses determined in Trial 232.
- Pharmacokinetics: To report delamanid and metabolite plasma concentrations at each visit by age groups and to conduct population pharmacokinetics (POPPK) anlaysis of delamanid when delamanid is administered in combination with an OBR during a 6-month treatment period in pediatric patients with MDR-TB.

#### 2.2 Secondary objectives:

- To evaluate the pharmacokinetic (PK)/ pharmacodynamics (PD) relationship of delamanid and its metabolite DM-6705 plasma concentrations and change in QTc when delamanid is administered in combination with OBR during a 6-month treatment period in pediatric patients with MDR-TB.
- Efficacy: To evaluate the efficacy of delamanid when administered in combination with an OBR during a 6-month treatment period in pediatric patients with MDR-TB.
- To determine the palatability of the delamanid pediatric formulation.

# 3 Study Design

This is a Phase 2, open-label, multi-dose, age de-escalation multicenter trial to assess the long-term safety, tolerability, PK, and efficacy of delamanid plus OBR over a 6-month treatment period in pediatric patients with MDR-TB who have successfully completed Trial 232. Since the trial is an extension of Trial 242-12-232 (Trial 232), patients must complete Trial 232 to roll-over to the current Trial 242-12-233 (Trial 233). Those patients who have completed Trial 232 and choose to enter Trial 233 must rollover from Trial 232 within 30 days after completing that Trial. If any patients terminate Trial 232 early or choose not to enter Trial 233, patients will be recruited to enter and complete Trial 232

first, and then rollover into Trial 233. However, patients who terminate Trial 233 early will not be replaced. Subject population is listed in Table 3-1 and study design schematic is illustrated in Figure 3-1.

Patients who enter Trial 233 will retain the same unique identification number and the same age group assigned to them in Trial 232:

| Table 3-1 | Subje | ect Population | |
|---|---|---|---|
| Group | Category | Sample Size (N) | Administration |
| 1† | Age 12 -17 years | 6+ | Adult formulation of delamanid 100 mg<br>BID + OBR for 6 months |
| 2‡ | Age 6 -11 years | 6+ | Adult formulation of delamanid 50 mg BID + OBR for 6 months |
| 3‡ | Age 3 -5 years | 12+ | Pediatric formulation of delamanid<br>(DPF) 25 mg BID + OBR for 6 months |
| 4* | Age 0 -2 years | 12+ | Pediatric formulation of delamanid based on body weight + OBR: Patient > 10 kg will receive DPF 10 mg BID + OBR Patient > 8 and <= 10 kg will receive DPF 5 mg BID + OBR Patient <= 8 kg will receive DPF 5 mg QD + OBR Delamanid dose will be adjusted as needed for Group 4 patients based on the weight measurement at specified study visits (Visits 5, 7, 9, 11 and 12) |

<sup>†</sup> Group 1 must include at least 2 but no more than 5 females.

Version Date: 3 July 2019

<sup>‡:</sup> Group 2, 3, 4 must include both genders.



Figure 3-1 Trial Design Schematic

# 4 Sample Size and Power Justification

Since patients are rolled over directly from Trial 232, no power/sample size calculation was performed for this trial and no formal statistical hypothesis test is planned due to the small sample size. All statistical presentations will be descriptive.

# 5 Statistical Analysis

## 5.1 General Principles

All data processing, summarization and analyses will be performed using version of 9.4 or higher of SAS®-statistical software packages. Data will be presented in summary tables by age groups, and by study time points if applicable.

Without distinction, Descriptive Continuous Statistics will include the number of patients / observations (N), mean, standard deviation (SD), min and max by default; Descriptive Categorical Statistics will include frequency counts and percentages [n (%)]. The denominator for percentage calculations will be the total number of patients in the analysis sample, or the subset of the analysis sample if the analyses are restricted for the subset of the analysis sample only, as defined in section 5.2, unless specified otherwise. No formal statistical hypothesis testing will be performed.

When a measurement is repeated for the same visit, the last of repeat values will be used for production of summary tables. International System of Units (SI) will be applied for all analyses unless specified otherwise.

# 5.2 Datasets for Analysis

For safety and PK summaries, the following study samples are defined in Analysis Data Model [ADaM] subject-level analysis dataset [ADSL] and naming conventions will follow Clinical Data Interchange Standards Consortium [CDISC] standards.

- Safety Sample: comprises the patients who have received any amount of study medication in Trial 233, regardless of any protocol deviation or violation.
- Efficacy Sample: comprises all patients with at least one efficacy endpoint available, the efficacy end points include: 1) chest radiograph result; 2) investigator assessed clinical signs and symptoms of tuberculosis; 3) microbiologic assessment of sputum; 4) evaluable change from baseline in body weight or height at treatment period.

#### 5.3 Definition of Baselines

Baseline is in general defined as the latest evaluation prior to the first dose in study 233, from both scheduled and unscheduled visits in either Trial 233, or Trial 232 if not applicable from Trial 233.

### 5.4 Handling of Missing Data

All analyses are performed on the observed data and no missing data imputation is needed.

## 5.5 Demographic and Baseline Characteristics

Baseline demographic characteristics including age, gender, race, ethnicity, height, height percentile for age, weight, weight percentile for age, body mass index (BMI) and menstruation will be summarized by age group for the Safety and Efficacy samples respectively using the baseline assessments. Descriptive statistics will be tabulated by age groups.

# 5.6 Medical History

General medical history will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) Version 18.0 (or a later version if updated during the study). All medical history will be listed, and Descriptive Categorical Statistics for patients with any medical history will be tabulated for safety sample by system organ class (SOC) and preferred term (PT) by age groups.

#### 5.7 Primary Outcome Analysis

# 5.7.1 Safety Outcome Variables

Safety and Tolerability was assessed by adverse events (AEs), physical examination including visual and audiometry assessments, vital signs, electrocardiograms, clinical laboratory tests (serum chemistry, hematology, urinalysis and other laboratory tests), .

Safety parameters will be summarized by incidence rates and their change from baseline if applicable. Change from baseline is summarized for observed cases at each scheduled post-baseline visit and for the last visit.

#### 5.7.1.1 Adverse Events

All adverse events (AEs) recorded will be classified by SOC and PT according to the most recent version of the Medical Dictionary for Regulatory Activities (MedDRA) available at the time of analysis.

Treatment emergent AE (TEAE) is defined as any new adverse event experienced by a study subject that occurs after the initiation of (investigational) Medicinal Product ((I)MP) administration; an event or pre-existing medical problem that has changed adversely in nature or severity from baseline in a patient/subject while receiving (I)MP.

The seriousness of AEs is assessed as "Death", "Life-threatening condition", "Persistent or significant incapacity", "Hospitalization- initial or prolonged", "Congenital anomaly or birth defect", "Medically significant condition" and "Non-serious".

The severity of all AEs is recorded as "Mild", "Moderate" and "Severe".

The relationship between an AE and study drug is assessed as "Related", "Possibly Related", "Unlikely Related" and "Not Related".

Action taken for AEs is recorded as "Drug Interrupted", "Drug Withdrawn", "Dose Not Changed", "Not Applicable" and "Unknown".

Adverse event outcome is assessed as "Recovered/Resolved", "Recovering/Resolving", "Recovered/Resolved with sequelae", "Not recovered/Not resolved", "Fatal" and "Unknown".

The number and percentage of the TEAEs will be summarized overall by SOC (sorted alphabetically) and PT (sorted by descending overall total).

Patients with more than one AE within a particular SOC or PT are counted only once for that PT and the maximum severity will be selected. AEs with missing intensity/severity

will be included in the overall count of patients with AEs, but will not be included in the counts in summary for severity.

- Incidence of TEAEs
- Incidence of TEAEs by severity
- Incidence of potentially drug-related TEAEs (including 'related' and 'possibly related')
- Incidence of TEAEs with an outcome of death
- Incidence of treatment-emergent serious adverse events
- Incidence of drug-discontinuations (drug withdrawn) due to TEAEs
- Incidence of non-serious AEs [NSAE] with incidence rate 5% or higher by System Organ Class and MedDRA Preferred Term.

#### 5.7.1.2 Clinical Laboratory Data

Data for the hematology, blood chemistry and urinalysis analytes received will be analyzed. The quantitative change in hematology, blood chemistry, and urinalysis analytes assessment results will be calculated relative to baseline. Laboratory tests with character results that cannot be quantitated by change from baseline will presented in tables with counts and percentages. Data obtained in the eCRF for additional analytes not required by the protocol will not be summarized, but will be included in listings.

Shift tables will be produced for assessing changes from baseline in clinical laboratory measurements using an ordinal scale (ie, low, normal, high based on lab normal range criteria).

Summary for frequency and percentage of laboratory tests that are newly occurred clinical significant during the study will be summarized for each laboratory parameter by age group. The clinical significant lab test result criteria is based on Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events[1]. Lab results with severity grade 3 or above is defined as clinical significant for this study and the criteria are listed in Appendix 1.

Listings of lab test results that are clinically significant will be presented.

A listing of all patients' lab result will be presented for each lab test and the values that are abnormal will be flagged as low (L) or high (H) in data listings.

If there are repeats for a certain lab test at a visit, then the last repeat value will be used in summaries. Post-baseline data from all unscheduled visits will not be included in the

Version Date: 3 July 2019

summary tables by visits, but will be included in clinical notable change table and listings.

# 5.7.1.3 Drug Induced Liver Injury (DILI)

The potential DILI case will be presented in tables and listings:

• AST or ALT  $\geq$  3 x ULN and total bilirubin to  $\geq$  2 ULN

#### 5.7.1.4 Physical Examination and Vital Signs

Vital signs will be listed and summarized by age groups and by visits:

- Weight (kg);
- Weight percentile for age.
- Height (cm);
- Height percentile for age
- Body temperature (°C);
- Heart rate (beats/min);
- Respiratory rate (breaths/minute);
- Systolic and diastolic blood pressure (mm Hg);
- BMI (kg/m2).

Physical examination [HEENT; Thorax; Abdomen; Urogenital; Extremities; Neurological; Skin and Mucosae] and vital signs data and changes from baseline in vital signs will be summarized by age group using Descriptive Continuous Statistics.

In addition, a listing of patients with at least one potentially clinically significant vital signs result will be presented for each vital sign parameter. Criteria for potentially clinically significant vital sign abnormalities are listed in Appendix 2. Summary for potentially clinically significant vital signs by visit, and newly acquired potentially clinically significant result during the treatment period will be presented for each vital sign by age group.

Post-baseline data from all unscheduled visits will not be included in the summary tables by visits, but will be included in clinical notable change table and listings.

# 5.7.1.5 Electrocardiogram Results

Continuous ECG parameters, including Heart rate, PR interval, QRS interval, QT intervals and QTc (including both QTcB and QTcF) will be summarized for:

• Descriptive Continuous Statistics on actual measurements and change from baseline.

• Summary table for patients with potentially clinically significant results. Criteria for potentially clinically significant vital sign abnormalities are listed in Appendix 3.

- Number and percentage of subjects with new qualitative abnormalities in rate, rhythm, conduction, morphology, including myocardial infarction, ST Segment, T Wave or U Wave abnormalities.
- Listing of patients with at least one potentially clinically significant ECG abnormalities result during the treatment period.

Data from all unscheduled visits will not be included in the summary tables for the changes from baseline by visits, but will be included in summary tables for the incidence of potentially clinically significant abnormalities and all listings.

#### 5.7.1.6 Additional Safety Assessments

Visual and audiometry assessment results will be summarized and listed by study visits.

#### 5.8 Extent of Exposure to Trial Medication

Number of days patients were exposed to IMP will be summarized by duration categories using counts and frequencies for the Safety Sample.

Duration of exposure to study drug will be defined as (date of last dose - date of first dose +1).

#### 5.9 Treatment Compliance

Acceptability of delamanid will be summarized by visit by age group. And the dose administration of delamanid will be listed and DOT plan compliance is shown in the listing.

#### 5.10 Protocol Deviation

Protocol deviations, as a measure of quality of study conduct, are summarized by type of deviation, and by age group for the safety sample, using Descriptive Categorical Statistics. Protocol deviations collected from CRF and generated from programmable cross-checks of data will be pooled together and listed by type of deviation, and by patient respectively. Nature of the violation, specified as either major or minor, will be included in the listing.

#### 5.11 Pharmacokinetic Analysis of Plasma

Delamanid and metabolite plasma concentrations will be reported with descriptive statistics at each visit day per age group. In addition, delamanid data from this trial will

be combined with PK data from Trial 232 for a separate population PK analysis and report and will be conducted by Clinical Pharmacology group.

### 5.11.1 Pharmacokinetic Assessment of Cerebral Spinal Fluid (CSF)

In patients where a lumbar puncture is clinically indicated during the routine management of a child enrolled in the trial, CSF concentrations of delamanid will be measured and reported. The delamanid CSF concentration will be listed by patient together with the timing of the lumbar puncture in relation to the timing of the dose. If adequate data is available, the concentrations will be summarized using descriptive statistics.

# 5.12 Secondary Outcome Analysis

#### 5.12.1 Pharmacokinetics/Phamacodynamics

PK/PD analysis will be performed by Clinical Pharmacology group to determine the relationship of delamanid and DM-6705 plasma concentrations any changes in QTc interval.

# 5.12.2 Efficacy Outcome Analysis

Descriptive Categorical Statistic will be summarized for each efficacy endpoint and presented in listings by patient, no formal statistical inference performed.

- Chest radiography results;
- Body weight/height
- Investigator-assessed signs and symptoms of tuberculosis:
  - 1) Cough;
  - 2) Fever;
  - 3) Weight loss;
  - 4) Failure to thrive;
  - 5) Hemoptysis;
  - 6) Dyspnea;
  - 7) Chest pain;
  - 8) Night sweats;
  - 9) Loss of appetite;
- Sputum culture conversion (SCC) will be assessed in patients with culture-positive and able to produce sputum or provide other biological specimens or with investigator order for purpose of routine management of the patient;

#### 5.12.3 Palatibility

The palatability of the pediatric formulation will be assessed using an age-appropriate visual hedonic scale and clinical assessment (Group 3 and 4 only). The counts and percentages will be tabulated in frequency tables.

# 5.12.4 Final Treatment Outcomes Assessed by the Principal Investigator

Final treatment outcomes will be assessed by the investigator at 24 months of initial IMP dose, according to the WHO outcome definitions for treating patients with MDR TB. Treatment outcome (Cured, Treatment Completed, Died, Treatment Failed, Lost to follow-up, Not evaluated) will be provided by treatment group. Frequency and percentage of patients achieving a favorable treatment outcome (cured or treatment completed) will be summarized by age group, using descriptive categorical statistics. Listing of treatment outcome will also be provided by age group.

#### 5.13 Concomitant Medications

Medications received concomitantly with study drug will be collected in the database and coded using the most recent WHO Drug Dictionary, Anatomical Therapeutic Chemical (ATC) Classification codes.

Descriptive Categorical Statistics will be tabulated by drug classification according to age group for the following periods:

- Prior to taking trial therapy;
- During the trial therapy;
- During the scheduled follow-up period after trial therapy complete.

# 5.14 Patient Disposition, Completion Rate and Reasons for Discontinuation

The number and percentage of patients who complete the trial and who discontinue early, including a breakdown of the primary reasons for discontinuation, will be summarized using Descriptive Categorical Statistics. Patients who are evaluated at the last scheduled visit of the trial, the follow-up visit (Visit 19, Day 365), will be defined as trial completers. The discontinuation by primary reasons will be summarized by age group for Enrolled and PK samples.

#### 5.15 Discontinuation

A patient disposition table will be presented including the following categories:

Safety (Treated)

Efficacy

PK

Early discontinued

Completed study treatment

The number and percentage of patients who complete the trial and who discontinue early, including a breakdown of the primary reasons for discontinuation, will be summarized using Descriptive Categorical Statistics. The discontinuation by primary reasons will be summarized by age group for Enrolled and PK samples:

Lost to follow-up

Adverse events

Sponsor discontinued study

Subject met withdrawal criteria

Subject was withdrawn from participation by the investigator

Subject withdrew consent to participate

Protocol deviation

# 5.16 Interim Analysis

Safety, tolerability, PK, and efficacy of delamanid in children 6 to 17 years of age will be reviewed when a full complete data is available.

# 6 Table of Contents for Table and Listings

- CT-1 PATIENT DISPOSITION ENROLLED SAMPLE
- CT-2 REASONS FOR DISCONTINUATION ENROLLED SAMPLE
- CT-3.1 DEMOGRAPHIC CHARACTERISTICS: AGE, WEIGHT, HEIGHT, BMI, GENDER, ETHNICITY, RACE AND COUNTRY SAFETY SAMPLE
- CT-3.2.1 AUDIOMETRY, CHEST X-RAY, AND VISUAL ASSESSMENT AT BASELINE SAFETY SAMPLE
- CT-3.2.2 INVESTIGATOR-ASSESSED SIGNS AND SYMPTOMS OF TUBERCULOSIS AT BASELINE SAFETY SAMPLE
- CT-3.2.3 ANTI-TB TREATMENT HISTORY SAFETY SAMPLE
- CT-3.2.4 SUMMARY OF MEDICAL HISTORY SAFETY SAMPLE
- CT-4.1.1 CONCOMITANT MEDICATIONS (EXCLUDING ANTI-TB MEDICATIONS): MEDICATIONS TAKEN PRIOR TO START OF TRIAL THERAPY SAFETY SAMPLE
- CT-4.1.2 CONCOMITANT MEDICATIONS(EXCLUDING ANTI-TB MEDICATIONS): MEDICATIONS TAKEN DURING STUDY THERAPY SAFETY SAMPLE
- CT-4.1.3 CONCOMITANT MEDICATIONS (EXCLUDING ANTI-TB MEDICATIONS): MEDICATIONS TAKEN AFTER END OF STUDY THERAPY SAFETY SAMPLE
- CT-4.2.1 CONCOMITANT ANTI-TB MEDICATIONS: MEDICATIONS TAKEN PRIOR TO START OF TRIAL THERAPY SAFETY SAMPLE
- CT-4.2.2 CONCOMITANT ANTI-TB MEDICATIONS: MEDICATIONS TAKEN DURING STUDY THERAPY SAFETY SAMPLE
- CT-4.2.3 CONCOMITANT ANTI-TB MEDICATIONS: MEDICATIONS TAKEN AFTER END OF STUDY THERAPY SAFETY SAMPLE
- CT-5.1 PHARMACOKINETIC PARAMETERS SAFETY SAMPLE
- CT-5.2 SUMMARY OF FINAL OUTCOME AT THE END OF TREATMENT AS ASSESSED BY PRINCIPAL INVESTIGATOR AT 24 MONTHS SAFETY SAMPLE
- CT-5.3 SUMMARY OF PALATABILITY OF DELAMINID SAFETY SAMPLE

- CT-5.4 SUMMARY OF AUDIOMETRY, CHEST X-RAY, AND VISUAL ASSESSMENTS SAFETY SAMPLE
- CT-5.5 SUMMARY OF INVESTIGATOR-ASSESSED SIGNS AND SYMPTOMS OF TUBERCULOSIS SAFETY SAMPLE
- CT-5.6 SUMMARY OF PERCENTILE OF WEIGHT AND HEIGHT SAFETY SAMPLE
- CT-6.1 PHARMACODYNAMIC ENDPOINTS SAFETY SAMPLE
- CT-6.2 LISTING OF CORRECTED QT INTERVALS AND PK PARAMETERS BY VISIT SAFETY SAMPLE
- CT-7.1 EXTENT OF EXPOSURE TO STUDY MEDICATION SAFETY SAMPLE
- CT-7.2 ADHERENCE TO STUDY MEDICATION SAFETY SAMPLE
- CT-8.1 ADVERSE EVENTS (ALL CAUSALITIES) SAFETY SAMPLE
- CT-8.2.1 INCIDENCE OF ALL TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS SAFETY SAMPLE
- CT-8.2.2 INCIDENCE OF ALL TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND MEDDRA PREFERRED TERM SAFETY SAMPLE
- CT-8.2.3 INCIDENCE OF ALL TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS, MEDDRA PREFERRED TERM AND SEVERITY SAFETY SAMPLE
- CT-8.3.1 INCIDENCE OF POTENTIALLY DRUG-RELATED TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS SAFETY SAMPLE
- CT-8.3.2 INCIDENCE OF POTENTIALLY DRUG-RELATED TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND MEDDRA PREFERRED TERM SAFETY SAMPLE
- CT-8.3.3 INCIDENCE OF POTENTIALLY DRUG-RELATED TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS, MEDDRA PREFERRED TERM AND SEVERITY SAFETY SAMPLE
- CT-8.4.1 INCIDENCE OF DEATH DUE TO TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS SAFETY SAMPLE

- CT-8.4.2 INCIDENCE OF DEATH DUE TO TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND MEDDRA PREFERRED TERM SAFETY SAMPLE
- CT-8.4.3 INCIDENCE OF DEATH BY SYSTEM ORGAN CLASS, MEDDRA PREFERRED TERM AND SEVERITY SAFETY SAMPLE
- CT-8.5.1 INCIDENCE OF SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS SAFETY SAMPLE
- CT-8.5.2 INCIDENCE OF SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND MEDDRA PREFERRED TERM SAFETY SAMPLE
- CT-8.5.3 INCIDENCE OF SERIOUS TREATMENT-EMERGENT ADVERSE EVENTS BY SYSTEM ORGAN CLASS, MEDDRA PREFERRED TERM AND SEVERITY SAFETY SAMPLE
- CT-8.6.1 INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS
  RESULTING IN DISCONTINUATION FROM STUDY MEDICATION BY SYSTEM
  ORGAN CLASS SAFETY SAMPLE
- CT-8.6.2 INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS
  RESULTING IN DISCONTINUATION FROM STUDY MEDICATION BY MEDDRA
  PREFERRED TERM SAFETY SAMPLE
- CT-8.6.3 INCIDENCE OF TREATMENT-EMERGENT ADVERSE EVENTS
  RESULTING IN DISCONTINUATION FROM STUDY MEDICATION BY MEDDRA
  PREFERRED TERM AND SEVERITY SAFETY SAMPLE
- CT-8.7.1 INCIDENCE (> 5%) OF NON-SERIOUS ADVERSE EVENTS BY SYSTEM ORGAN CLASS AND MEDDRA PREFERRED TERM SAFETY SAMPLE
- CT-8.8.1 LISTING OF DEATHS SAFETY SAMPLE
- CT-8.8.2 LISTING OF SERIOUS ADVERSE EVENTS SAFETY SAMPLE
- CT-8.8.3 LISTING OF DISCONTINUATIONS DUE TO ADVERSE EVENTS SAFETY SAMPLE
- CT-9 SUMMARY OF PHYSICAL EXAMINATION SAFETY SAMPLE
- CT-10.1.1 MEAN CHANGE FROM BASELINE IN LABORATORY TEST RESULTS: SERUM CHEMISTRY SAFETY SAMPLE

CT-10.1.2 MEAN CHANGE FROM BASELINE IN LABORATORY TEST

RESULTS: HEMATOLOGY SAFETY SAMPLE

CT-10.1.3 MEAN CHANGE FROM BASELINE IN LABORATORY TEST

RESULTS: URINALYSIS SAFETY SAMPLE

CT-10.1.4 MEAN CHANGE FROM BASELINE IN LABORATORY TEST

RESULTS: OTHERS SAFETY SAMPLE

CT-10.1.5 SUMMARY OF CATEGORICAL LABORATORY TEST RESULTS:

URINALYSIS SAFETY SAMPLE

CT-10.2.1 SHIFT TABLES OF CLINICAL LABORATORY TEST RESULTS:

SERUM CHEMISTRY SAFETY SAMPLE

CT-10.2.2 SHIFT TABLES OF CLINICAL LABORATORY TEST RESULTS:

HEMATOLOGY SAFETY SAMPLE

CT-10.2.3 SHIFT TABLES OF CLINICAL LABORATORY TEST RESULTS:

URINALYSIS SAFETY SAMPLE

CT-10.2.4 SHIFT TABLES OF CLINICAL LABORATORY TEST RESULTS:

OTHERS SAFETY SAMPLE

CT-10.3.1 LISTING OF LABORATORY TEST VALUES OUTSIDE NORMAL

RANGES, BY AGE GROUP: SERUM CHEMISTRY SAFETY SAMPLE

CT-10.3.2 LISTING OF LABORATORY TEST VALUES OUTSIDE NORMAL

RANGES, BY AGE GROUP: HEMATOLOGY SAFETY SAMPLE

CT-10.3.3 LISTING OF LABORATORY TEST VALUES OUTSIDE NORMAL

RANGES, BY AGE GROUP: URINALYSIS SAFETY SAMPLE

CT-10.3.4 LISTING OF LABORATORY TEST VALUES OUTSIDE NORMAL

RANGES, BY AGE GROUP: OTHERS SAFETY SAMPLE

CT-10.3.5 CRITERIA FOR LABORATORY TEST VALUES OUTSIDE NORMAL

RANGES SAFETY SAMPLE

CT-10.4.1 INCIDENCE OF CLINICALLY SIGNIFICANT LABORATORY TEST

ABNORMALITIES: SERUM CHEMISTRY SAFETY SAMPLE

CT-10.4.2 INCIDENCE OF CLINICALLY SIGNIFICANT LABORATORY TEST

ABNORMALITIES: HEMATOLOGY SAFETY SAMPLE

CT-10.4.3 INCIDENCE OF CLINICALLY SIGNIFICANT LABORATORY TEST ABNORMALITIES: URINANALYSIS SAFETY SAMPLE

CT-10.5.1 INCIDENCE OF NEWLY ACQUIRED CLINICALLY SIGNIFICANT LABORATORY TEST ABNORMALITIES FROM BASELINE: SERUM CHEMISTRY SAFETY SAMPLE

CT-10.5.2 INCIDENCE OF NEWLY ACQUIRED CLINICALLY SIGNIFICANT LABORATORY TEST ABNORMALITIES FROM BASELINE: HEMATOLOGY SAFETY SAMPLE

CT-10.5.3 INCIDENCE OF NEWLY ACQUIRED CLINICALLY SIGNIFICANT LABORATORY TEST ABNORMALITIES FROM BASELINE: URINANALYSIS SAFETY SAMPLE

CT-10.5.4 CRITERIA FOR POTENTIALLY CLINICAL SIGNIFICANT LABORATORY TEST ABNORMALITIES SAFETY SAMPLE

CT-10.6.1 LISTING OF CLINICALLY SIGNIFICANT LABORATORY ABNORMALITIES: SERUM CHEMISTRY SAFETY SAMPLE

CT-10.6.2 LISTING OF CLINICALLY SIGNIFICANT LABORATORY ABNORMALITIES: HEMATOLOGY SAFETY SAMPLE

CT-10.6.3 LISTING OF CLINICALLY SIGNIFICANT LABORATORY ABNORMALITIES: URINANALYSIS SAFETY SAMPLE

CT-10.7.1 INCIDENCE AND PERCENTAGE OF ELEVATED LIVER ENZYMES AND POTENTIAL DRUG INDUCED LIVER INJURY SAFETY SAMPLE

CT-10.7.2 LISTING OF AST OR ALT  $\ge$  3 x ULN WITH  $\ge$  2 x ULN IN BILIRUBIN SAFETY SAMPLE

CT-11.1 MEAN CHANGE FROM BASELINE IN VITAL SIGN PARAMETERS SAFETY SAMPLE

CT-11.2 INCIDENCE OF CLINICALLY SIGNIFICANT ABNORMALITY IN VITAL SIGN SAFETY SAMPLE

CT-11.3 LISTING OF POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITY IN VITAL SIGNS SAFETY SAMPLE

CT-11.4 CRITERIA FOR POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITY IN VITAL SIGNS SAFETY SAMPLE

CT-12.1 MEAN CHANGE FROM BASELINE IN ELECTROCARDIOGRAM PARAMETERS SAFETY SAMPLE

CT-12.2 INCIDENCE OF CLINICALLY SIGNIFICANT ELECTROCARDIOGRAM TEST ABNORMALITIES SAFETY SAMPLE

CT-12.3 LISTING OF POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITY IN ELECTROCARDIOGRAM SAFETY SAMPLE

CT-12.4 CRITERIA FOR POTENTIALLY CLINICALLY SIGNIFICANT ABNORMALITY IN ELECTROCARDIOGRAM SAFETY SAMPLE

PDATA-1 ENTRANCE CRITERIA

PDATA-2 ELIGIBILITY: INCLUSION-EXCLUSION CRITERIA

PDATA-3.1 SUBJECT DISPOSITION

PDATA-3.2 STUDY COMPLETION STATUS AND REASONS FOR DISCONTINUATION

PDATA-4.1 DEMOGRAPHIC CHARACTERISTICS: AGE, SEX, HEIGHT, WEIGHT, BMI, RACE, AND ETHNICITY

PDATA-4.2 AUDIOMETRY, CHEST X-RAY, AND VISUAL ASSESSMENTS

PDATA-4.3 INVESTIGATOR-ASSESSED SIGNS AND SYMPTOMS OF TUBERCULOSIS

PDATA-4.4 PREGNANCY TEST RESULTS

PDATA-4.5 SPECIMEN COLLECTION FOR MICROBIOLOGY TEST RESULTS

PDATA-4.6 PALATABILITY ASSESSMENT

PDATA-5 GENERAL MEDICAL HISTORY

PDATA-6.1 CONCOMITANT MEDICATIONS: MEDICATIONS TAKEN PRIOR TO START OF STUDY THERAPY

PDATA-6.2 CONCOMITANT MEDICATIONS: MEDICATIONS TAKEN DURING STUDY THERAPY

PDATA-6.3 CONCOMITANT MEDICATIONS: MEDICATIONS TAKEN AFTER END OF STUDY THERAPY

PDATA-6.4 CONCOMITANT ANTI-TB MEDICATIONS: MEDICATIONS TAKEN PRIOR TO START OF STUDY THERAPY

PDATA-6.5 CONCOMITANT ANTI-TB MEDICATIONS: MEDICATIONS TAKEN DURING STUDY THERAPY

PDATA-6.6 CONCOMITANT ANTI-TB MEDICATIONS: MEDICATIONS TAKEN AFTER END OF STUDY THERAPY

PDATA-7.1 DOSE ADMINISTRATION

PDATA-7.2 STUDY MEDICATION

PDATA-7.3 STUDY MEDICATION ACCOUNTABILITY

PDATA-7.4 OBR ACCEPTABILITY

PDATA-8.1 PHYSICAL EXAMINATION

PDATA-8.2 MENSTRUATION

PDATA-9 VITAL SIGNS

PDATA-10.1 ELECTROCARDIOGRAM RESULTS

PDATA-10.2 ELECTROCARDIOGRAM RESULTS - DIAGNOSIS

PDATA-11 ADVERSE EVENTS

PDATA-12 PK BLOOD SAMPLING

PDATA-13 LAST DOSE OF DELAMANID PRIOR TO PK SAMPLING

PDATA-14 LISTING OF TUBERCULOSIS DIAGNOSIS RESULT

PDATA-15 TREATMENT OUTCOME

DEMOG-1 LISTING OF DEMOGRAPHIC CHARACTERISTICS

DREAS-1 DISCONTINUED SUBJECTS AND REASON FOR DISCONTINUATION

SMED-1 STUDY MEDICATION COMPLIANCE OF OPC-67683

AE-1 ADVERSE EVENTS

LAB-1 LABORATORY TEST RESULTS: SERUM CHEMISTRY

LAB-2 LABORATORY TEST RESULTS: HEMATOLOGY

LAB-3 LABORATORY TEST RESULTS: URINALYSIS

LAB-4 LABORATORY TEST RESULTS: OTHERS

PDEV-1 SUMMARY OF PROTOCOL DEVIATIONS BY AGE GROUP AND TYPE OF DEVIATION

- PDEV-2 PROTOCOL DEVIATIONS BY DEVIATION TYPE
- PDEV-3 LISTING OF PROTOCOL DEVIATIONS
- PDEV-4 PROTOCOL DEVIATIONS CRITERIA

# 7 Bibliography

1 Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events. Version 2.1. July 2017

Appendix 1 Serum Chemistry, Hematology and Urinalysis Lab Test Results Clinical Significant Criteria Based on Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events

| LAB GROUP | TEST | UNITS | SEX | AGE Group | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|---|---|
| Chemistry | Albumin, Low | g/dL | Male/Female | All | < 2.0 | NA |
| Chemistry | Albumin, Low | g/L | Male/Female | All | < 20 | NA |
| Chemistry | Alkaline Phosphatase, High | | Male/Female | All | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Chemistry | ALT or SGPT, High | | Male/Female | All | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Chemistry | AST or SGOT, High | | Male/Female | All | 5.0 to < 10.0 x ULN | ≥ 10.0 x ULN |
| Chemistry | Total Bilirubin, High | | Male/Female | > 28 days of age | 2.6 to < 5.0 x ULN | ≥ 5.0 x ULN |
| Chemistry | Calcium, High | mg/dL | Male/Female | ≥ 7 days of age | 12.5 to < 13.5 | ≥ 13.5 |
| Chemistry | Calcium, High | mmol/L | Male/Female | ≥ 7 days of age | 3.13 to < 3.38 | ≥ 3.38 |
| Chemistry | Calcium, Low | mg/dL | Male/Female | ≥ 7 days of age | 6.1 to < 7.0 | < 6.1 |
| Chemistry | Calcium, Low | mmol/L | Male/Female | ≥ 7 days of age | 1.53 to < 1.75 | < 1.53 |
| Chemistry | Creatinine, High | | Male/Female | All | > 1.8 to $< 3.5$ x ULN | ≥ 3.5 x ULN |
| Chemistry | Glucose, High | mg/dL | Male/Female | All | > 250 to 500 | ≥ 500 |
| Chemistry | Glucose, High | mmol/L | Male/Female | All | 13.89 to < 27.75 | ≥ 27.75 |
| Chemistry | Glucose, Low | mg/dL | Male/Female | $\geq 1$ month of age | 30 to < 40 | < 30 |
| Chemistry | Glucose, Low | mmol/L | Male/Female | $\geq 1$ month of age | 1.67 to < 2.22 | < 1.67 |
| Chemistry | Cholesterol, High | mg/dL | Male/Female | All | ≥ 300 | NA |
| Chemistry | Cholesterol, High | mmol/L | Male/Female | All | ≥ 7.77 | NA |
| Chemistry | Inorganic Phosphorus, Low | mg/dL | Male/Female | > 14 years of age | 1.0 to < 1.4 | < 1.0 |
| Chemistry | Inorganic Phosphorus, Low | mmol/L | Male/Female | > 14 years of age | 0.32 to < 0.45 | < 0.32 |
| Chemistry | Inorganic Phosphorus, Low | mg/dL | Male/Female | <1 to 14 years of age | 1.5 to < 2.5 | < 1.5 |
| Chemistry | Inorganic Phosphorus, Low | mmol/L | Male/Female | <1 to 14 years of age | 0.48 to < 0.81 | < 0.48 |
| Chemistry | Magnesium, Low | mEq/L | Male/Female | All | 0.6 to < 0.9 | < 0.6 |
| Chemistry | Magnesium, Low | mmol/L | Male/Female | All | 0.30 to < 0.45 | < 0.30 |
| Chemistry | Potassium, High | mEq/L | Male/Female | All | 6.5 to < 7.0 | ≥ 7.0 |
| Chemistry | Potassium, High | mmol/L | Male/Female | All | 6.5 to < 7.0 | ≥ 7.0 |

| LAB GROUP | TEST | UNITS | SEX | AGE Group | GRADE 3<br>SEVERE | GRADE 4<br>POTENTIALLY LIFE-<br>THREATENING |
|---|---|---|---|---|---|---|
| Chemistry | Potassium, Low | mEq/L | Male/Female | All | 2.0 to < 2.5 | < 2.0 |
| Chemistry | Potassium, Low | mmol/L | Male/Female | All | 2.0 to < 2.5 | < 2.0 |
| Chemistry | Sodium, High | mEq/L | Male/Female | All | 154 to < 160 | ≥ 160 |
| Chemistry | Sodium, High | mmol/L | Male/Female | All | 154 to < 160 | ≥ 160 |
| Chemistry | Sodium, Low | mEq/L | Male/Female | All | 121 to < 125 | ≤ 120 |
| Chemistry | Sodium, Low | mmol/L | Male/Female | All | 121 to < 125 | ≤ 120 |
| Chemistry | Triglycerides, High | mg/dL | Male/Female | All | >500 to < 1,000 | > 1,000 |
| Chemistry | Triglycerides, High | mmol/L | Male/Female | All | >5.7 to 11.4 | > 11.4 |
| Chemistry | Uric Acid, High | mg/dL | Male/Female | All | 12.0 to < 15.0 | ≥ 15.0 |
| Chemistry | Uric Acid, High | mmol/L | Male/Female | All | 0.71 to < 0.89 | $\geq 0.89$ |
| Hematology | Activated Partial Thromboplastin<br>Time, High | | Male/Female | All | 2.33 to < 3.00 x ULN | ≥ 3.00 x ULN |
| Hematology | Absolute CD4+ Count, Low | cell/mm <sup>3</sup> | Male/Female | All> 5 years of age (not HIV infected) | 100 to < 200 | < 100 |
| Hematology | Absolute CD4+ Count, Low | cells/L | Male/Female | > 5 years of age<br>(not HIV infected) | 100 to < 200 | < 100 |
| Hematology | Absolute Lymphocytes, Low | cell/mm <sup>3</sup> | Male/Female | > 5 years of age<br>(not HIV infected) | 350 to < 500 | < 350 |
| Hematology | Absolute Lymphocytes, Low | cells/L | Male/Female | > 5 years of age<br>(not HIV infected) | $0.350 \times 10^9 \text{ to} < 0.500 \times 10^9$ | < 0.350 x 10 <sup>9</sup> |
| Hematology | Absolute Neutrophil Count, Low | cell/mm <sup>3</sup> | Male/Female | > 7 days of age | 400 to 599 | <400 |
| Hematology | Absolute Neutrophil Count, Low | cells/L | Male/Female | > 7 days of age | $0.400 \times 10^9 \text{ to} < 0.599 \times 10^9$ | $< 0.400 \times 10^9$ |
| Hematology | Hemoglobin, Low | g/dL | Male | ≥ 13 years of age | 7.0 to < 9.0 | < 7.0 |
| Hematology | Hemoglobin, Low | mmol/L | Male | $\geq$ 13 years of age | 4.34 to < 5.57 | < 4.34 |
| Hematology | Hemoglobin, Low | g/dL | Female | ≥ 13 years of age | 6.5 to < 8.5 | < 6.5 |
| Hematology | Hemoglobin, Low | mmol/L | Female | $\geq$ 13 years of age | 4.03 to < 5.25 | < 4.03 |
| Hematology | Hemoglobin, Low | g/dL | Male/Female | 57 days of age to < 13 years of age | 6.5 to < 8.5 | < 6.5 |
| Hematology | Hemoglobin, Low | mmol/L | Male/Female | 57 days of age to < 13 years of age | 4.03 to < 5.25 | < 4.03 |
| Hematology | Platelet Count, Decreased | cells/mm <sup>3</sup> | Male/Female | All | 25,000 to < 50,000 | < 25,000 |
| Hematology | Platelet Count, Decreased | cells/L | Male/Female | All | 25.000 x 10 <sup>9</sup> to < 50.000 x 10 <sup>9</sup> | < 25.000 x 10 <sup>9</sup> |
| Hematology | Prothrombin Time, High | | Male/Female | All | 1.50 to < 3.00 x ULN | ≥ 3.00 x ULN |

| LAB GROUP | TEST | UNITS | SEX | AGE Group | GRADE 3<br>SEVERE | GRADE 4 POTENTIALLY LIFE- THREATENING |
|---|---|---|---|---|---|---|
| Hematology | Partial Thromboplastin Time, High | | Male/Female | All | 2.33 to < 3.00 x ULN | $\geq 3.00 \text{ x ULN}$ |
| Hematology | White Blood Cell, Decreased | cells/mm <sup>3</sup> | Male/Female | > 7 days of age | 1,000 to 1,499 | < 1,000 |
| Hematology | White Blood Cell, Decreased | cells/L | Male/Female | > 7 days of age | 1.000 x 10 <sup>9</sup> to 1.499 x 10 <sup>9</sup> | < 1.000 x 10 <sup>9</sup> |
| Urinalysis | Urine Glucose | | Male/Female | All | > 2+ or >500 mg | NA |
| Urinalysis | Urine Blood | | Male/Female | All | Gross OR Presence of RBC casts OR Intervention indicated | Life-threatening consequences |
| Urinalysis | Urine Protein | | Male/Female | All | 3+ or higher | NA |

RBC = red blood cell; ULN=upper normal limit

Appendix 2 Criteria for Potentially Clinical Significant Vital Sign Abnormalities

| Variable | Change Relative to Baseline |
|----------|---------------------------------|
| Weight | Decrease of >=5% in body weight |
| | Increase of >=5% in body weight |

Note: In order to be identified as "potentially clinical significant abnormal," an on-drug value must represent a change from the patient's baseline value of at least the magnitude shown in the "Change Relative to Baseline column.

Appendix 3 Criteria for Potentially Clinical Significant ECG
Abnormalities

| Classification | Criterion Value | Change Relative to Baseline |
|---|---|---|
| HR Outliers | < 50 bpm | Decrease of >= 25% |
| | > 100 bpm | Increase of >= 25% |
| PR Outliers | > 200 msec | Increase of >= 25% |
| QRS Outliers | > 100 msec | Increase of >= 25% |
| QT | New Onset (> 500 msec) § | |
| QTcB | New Onset (> 450 msec) §<br>New Onset (> 480 msec) § | Increase of >= 30 msec and <=60 msec |
| | New Onset (> 500 msec) § | Increase of >60 msec |
| OTcF | New Onset (> 450 msec) §<br>New Onset (> 480 msec) § | Increase of >= 30 msec and <=60 msec |
| | New Onset (> 500 msec) § | Increase of > 60 msec |
| U Waves | New Abnormal U Waves | |
| ST Segment | New ST Segment Changes | |
| T Waves | New T Wave Changes | |
| Rhythm | New Abnormal Rhythm | |
| Conduction | New Conduction Abnormality | |

Note: In order to be identified as "potentially clinical significant abnormal," an on-drug value must meet the "Criterion Value" and also represent a change from the patient's pretreatment value of at least the magnitude shown in the "Change Relative to Baseline column.

<sup>§</sup> New Onset is defined as "not present on baseline ECG but present on on-treatment ECG". New Onset (> 450 msec), or New Onset (> 480 msec), or New Onset (> 500 msec) means a patient who attains a value >450 msec, or >480 msec, >500 msec respectively during treatment period but not at baseline visit.



# This page is a manifestation of an electronically captured signature

# SIGNATURE PAGE

Document Name: SAP-242-12-233

Document Number: 1000044284

**Document Version: 2.0** 

| Signed by | Meaning of Signature | Server Date (dd-MMM- yyyyy hh:min) - UTC timezone |
|---|---|---|
| | Biostatistics Approval | 03-Jul-2019<br>16:25:04 |
| | Clinical Pharmacology<br>Approval | 08-Jul-2019<br>14:58:26 |
| | Clinical Approval | 03-Jul-2019<br>18:56:36 |